CLINICAL TRIAL: NCT05851222
Title: Predicting Acute Kidney Injury in Infants Exposed to Nephrotoxic Drugs: A Big Data Approach to Predict NEOnatal Acute Kidney Injury in Newborns expoSed to nephroTOxic Drugs. (NeoAKI STOP)
Brief Title: A Big Data Approach to Predict NEOnatal Acute Kidney Injury in Newborns expoSed to nephroTOxic Drugs (NeoAKI STOP)
Acronym: NeoAKISTOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Giacomo Cavallaro, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: NeoAKI STOP
Record Dates: First submitted 2023-04-09; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Acute Kidney Injury; Drug Use; Drug Interaction; Drug Toxicity; Drug-Induced Nephropathy; Machine Learning; Newborn Morbidity; Premature Birth
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational retrospective study aims to learn about the incidence of acute kidney (AKI) injury in newborns in infants exposed to nephrotoxic drugs with a big data approach.

The main question it aims to answer are:

* Develop a model that can predict the occurrence of AKI in infants admitted to the NICU;
* Identify the drug or combination of drugs associated with an increased risk of AKI.

The group of infants exposed to drugs will be defined based on exposure for at least 1-day tone one or more therapies commonly used in the NICU. Once the AKI event has occurred, the observation of the trend of daily creatinine and diuresis values will be continued for the period covered by the study.

DETAILED DESCRIPTION:
1. Rationale and background Acute Kidney Injury (AKI) is defined as the sudden impairment of kidney function that results in altered hydro electrolyte balance and renal waste product elimination.

   Extensive evidence shows that the onset of AKI in critically ill pediatric patients is associated with an increased risk of death and a longer length of hospitalization. Furthermore, in patients who survive an episode of AKI, there is an increased risk of developing long-term morbidity, particularly Chronic Kidney Disease (CKD).

   The neonatal kidney has numerous features on the pathophysiological level that predispose this population more to AKI than at other life ages.

   In addition to the peculiarities related to the development and physiology of the kidney, especially if preterm, infants admitted to the NICU are exposed to multiple risk factors that may contribute to the onset of AKI.

   A recent multicenter study conducted in neonatal intensive care units in Canada, Australia, India, and the United States reported an overall incidence of AKI of 29.9% and showed that the development of AKI is an independent risk factor for death and prolonged hospitalization. The incidence of AKI by gestational age also showed a typical U-shaped distribution, with the greater occurrence at the two extremes represented by infants with gestational ages >36 weeks (36.7%) and <29 weeks (47.9%), while the lowest value was recorded in the 29-36 weeks range.

   The risk of developing acute kidney injury is known to increase with the number of medications used (especially if > 3) and the duration of exposure, especially for the aminoglycoside antibiotic category. In addition, critically ill patients who developed AKI were generally more exposed to nephrotoxic drugs than those who did not develop AKI. In the NICU setting, it is estimated that 87% of VLBW infants are exposed to at least one nephrotoxic drug during their hospital stay, and about a quarter of these infants develop at least one episode of acute renal distress.

   The diagnosis of AKI is based on increased serum creatinine (SCr) or decreased urinary output.

   To date, the definition of acute kidney injury is based on the former Kidney Disease Improving Global Outcomes (KIDGO) criteria modified for newborns.

   However, in light of the premises made, it can be understood how creatinine monitoring allows only passive observation of the phenomenon, noting the rise in creatinine values when renal insult has already occurred by then. This allows only retrospective changes in some aspects of the infant's management, such as optimizing fluid intake, suspending the administration of nephrotoxic drugs, and correcting any electrolyte imbalances, but without being able to prevent the onset of AKI. Ideally, the investigators should be able to understand and predict how different risk factors contribute to the beginning of renal damage in a given patient, thus allowing individualized management.

   Given the complexity of patients admitted to the NICU and the number of variables in the field, the problem lends itself well to analysis through AI and general statistical inference methods. Such methods have previously been used successfully for studies on adult patients but, to our knowledge, never on newborn patients.

   The investigators hope to apply these models in a prospective cohort study to validate their use and develop a real-time monitoring system of the kidney well-being of our nephrotoxic drug-exposed infants that can guide the clinician in patient management. Indeed, systematic surveillance of at-risk patients can significantly reduce the onset of kidney damage and limit both short-term and long-term consequences, thereby improving neonatal outcomes.
2. Research question and objectives 2.1 Primary objectives

   * Develop a model that can predict the occurrence of AKI in infants admitted to the NICU;
   * Identify the drug or combination associated with an increased risk of AKI. 2.2 Secondary objectives
   * Identify subgroups of patients at increased risk of AKI;
   * Identify time windows at increased risk of AKI during NICU admission.
3. Methods 3.1 Study design Single-center retrospective observational cohort study at the UOC of Neonatology and Neonatal Intensive Care Unit of Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy.

   3.1.1 Primary endpoints

   • Development of AKI defined according to modified KIDGO criteria for the newborn based on increased serum creatinine values or reduced mean hourly diuresis during NICU admission.

   3.1.2 Secondary endpoints
   * Number of AKI cases in risk subcategories: very low birth weight (birth weight < 1500 g), extremely low birth weight (birth weight < 1000 g), cardiopathic, with surgical pathology, sepsis, asphyxia;
   * Number of AKI cases in the first week of hospitalization compared with other periods.
4. Setting A population of infants admitted to the NICU of the Foundation will be retrospectively considered.

   4.1 Study population The study population will consist of patients born between January 2010 and December 2022.
5. Inclusion criteria

   • Patients who meet all of the following criteria will be included in the study:
   * born between 01/01/2010 and 31/12/2022;
   * admitted within 24 hours of birth in the NICU (both inborn and outborn);
   * availability of at least two serum creatinine values or a daily hourly diuresis assessment in the first 30 days of life.
6. Exclusion Criteria

   Patients who meet even one of the following criteria will be excluded:
   * pre- or postnatal diagnosis of severe urologic and/or nephrologic pathology on a malformative and/or genetic basis;
   * finding of serum creatinine > 2 mg/dl in the first 24 hours of life;
   * genetic conditions that may impact patient survival or renal function;
   * length of stay in the NICU less than 48 hours (death or transfer to another department);
   * infants undergoing ECMO.
7. Variables Clinical and instrumental data regarding each patient's medical history will be acquired for the NICU admission by the first month of life.

   Definition of AKI All available serum creatinine values for each patient during the NICU admission will be recorded, considering that determinations made within the first 48 hours of the infant's life are affected by maternal creatinine values.

   The presence of AKI will be determined according to the modified KIDGO criteria for the newborn, as reported in previous work in the neonatal setting.

   Exposure to drugs. The group of infants exposed to drugs will be defined based on exposure for at least 1-day tone one or more therapies commonly used in the NICU. Special attention will be given to exposure to antibiotics, antivirals, antifungals, diuretics, anti-inflammatories, inotropes, and vasopressors. In addition to the active ingredient, other significant data such as prescribed dose, administration route, treatment duration, and temporal relationship between treatment and diagnosis of AKI will also be considered. Once the AKI event has occurred, the observation of the trend of daily creatinine and diuresis values will be continued for the period covered by the study.
8. Source documents Data will be collected from each newborn's Neocare electronic medical record (GPI SpA).
9. Sample size Approximately 600 newborns are admitted to the neonatal intensive care unit each year. The incidence of renal damage in the critically ill newborn population is reported in the literature to be approximately 30%. In light of these considerations, over the decade of our observation, the estimated number of infants admitted to the NICU is about 6000 patients. Assuming a 30% drop-out related to exclusion criteria (about 1800 subjects), the investigators expect to be able to include approximately 4200 subjects in the study, among whom the investigators should find about 1200 cases of acute renal damage.
10. Data management Data will be collected anonymously by assigning a code to each patient. They will then be organized and stored on data storage systems with secure access.
11. Data Analysis Data will be analyzed using statistical inference approaches peculiar to Data Science and Artificial Intelligence (AI), such as Decision Trees, Logistic Regression, and Machine Learning (ML). The data themselves will suggest the choice of methods used.
12. Primary endpoint: analysis Identifying patterns or items in the administration of so-called off-label drugs in the neonatal patient (premature or not) and the development of renal syndromes related to the administration of the drug itself. Once one or more correlation factors have been identified, they could be entered within the Electronic Medical Record system (and in particular within the Clinical Decision Support System) in order to be able to alert the treating clinical staff of any clinical risk associated with the administration.
13. Secondary endpoint: analysis Development of a computational Early Warning model for AKI that ensures the interpretability of the prediction.

ELIGIBILITY:
Inclusion Criteria:

* born between 01/01/2010 and 31/12/2022;
* admitted within 24 hours of birth in the NICU (both inborn and outborn);
* availability of at least two serum creatinine values or a daily hourly diuresis assessment in the first 30 days of life.

Exclusion Criteria:

* pre- or postnatal diagnosis of severe urologic and/or nephrologic pathology on a malformative and/or genetic basis;
* finding of serum creatinine > 2 mg/dl in the first 24 hours of life;
* genetic conditions that may impact patient survival or renal function;
* length of stay in the NICU less than 48 hours (death or transfer to another department);
* infants undergoing ECMO.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to NICU and born between January 2010 and December 2022
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop a model that can predict the occurrence of AKI in infants admitted to the NICU; | From the date of randomization until the date of the first documented progression of AKI and up to 4 weeks
  All available serum creatinine values for each patient during the NICU admission will be recorded, considering that determinations made within the first 48 hours of the infant's life are affected by maternal creatinine values.
  The presence of AKI will be determined according to the modified KIDGO criteria for the newborn, as reported in previous work in the neonatal setting (Jetton JG, 2017; Jetton JG and Askenazi DJ, 2012; Stoops C, 2016; Askenazi DJ, Patil NR, et al., 2015; Sarkar S, 2014).
Identify the drug or combination of drugs associated with an increased risk of AKI | From the date of randomization until the date of the first documented progression of AKI and up to 4 weeks
  The group of infants exposed to drugs will be defined based on exposure for at least 1-day tone one or more therapies commonly used in the NICU. Special attention will be given to exposure to antibiotics, antivirals, antifungals, diuretics, anti-inflammatories, inotropes, and vasopressors. In addition to the active ingredient, other significant data such as prescribed dose, administration route, treatment duration, and temporal relationship between treatment and diagnosis of AKI will also be considered.

SECONDARY OUTCOMES:
Identify subgroups of patients at increased risk of AKI | From the date of randomization until the date of the first documented progression of AKI and up to 4 weeks
  Number of AKI cases in risk subcategories: very low birth weight (birth weight < 1500 g), extremely low birth weight (birth weight < 1000 g), cardiopathic, with surgical pathology, sepsis, asphyxia
Identify time windows at increased risk of AKI during NICU admission. | From the date of randomization until the date of the first documented progression of AKI and up to 4 weeks
  Number of AKI cases in the first week of hospitalization compared with other periods

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Cavallaro, MD, PhD, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Ilaria Amodeo, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Neonatal Intensive Care Unit, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abitbol CL, Seeherunvong W, Galarza MG, Katsoufis C, Francoeur D, Defreitas M, Edwards-Richards A, Master Sankar Raj V, Chandar J, Duara S, Yasin S, Zilleruelo G. Neonatal kidney size and function in preterm infants: what is a true estimate of glomerular filtration rate? J Pediatr. 2014 May;164(5):1026-1031.e2. doi: 10.1016/j.jpeds.2014.01.044. Epub 2014 Mar 5. PMID 24607244
- [Result] Askenazi D, Patil NR, Ambalavanan N, Balena-Borneman J, Lozano DJ, Ramani M, Collins M, Griffin RL. Acute kidney injury is associated with bronchopulmonary dysplasia/mortality in premature infants. Pediatr Nephrol. 2015 Sep;30(9):1511-8. doi: 10.1007/s00467-015-3087-5. Epub 2015 Mar 26. PMID 25808019
- [Result] Askenazi DJ, Feig DI, Graham NM, Hui-Stickle S, Goldstein SL. 3-5 year longitudinal follow-up of pediatric patients after acute renal failure. Kidney Int. 2006 Jan;69(1):184-9. doi: 10.1038/sj.ki.5000032. PMID 16374442
- [Result] Askenazi DJ, Koralkar R, Hundley HE, Montesanti A, Parwar P, Sonjara S, Ambalavanan N. Urine biomarkers predict acute kidney injury in newborns. J Pediatr. 2012 Aug;161(2):270-5.e1. doi: 10.1016/j.jpeds.2012.02.007. Epub 2012 Mar 16. PMID 22424940
- [Result] Askenazi DJ, Koralkar R, Hundley HE, Montesanti A, Patil N, Ambalavanan N. Fluid overload and mortality are associated with acute kidney injury in sick near-term/term neonate. Pediatr Nephrol. 2013 Apr;28(4):661-6. doi: 10.1007/s00467-012-2369-4. Epub 2012 Dec 9. PMID 23224224
- [Result] Askenazi DJ, Koralkar R, Levitan EB, Goldstein SL, Devarajan P, Khandrika S, Mehta RL, Ambalavanan N. Baseline values of candidate urine acute kidney injury biomarkers vary by gestational age in premature infants. Pediatr Res. 2011 Sep;70(3):302-6. doi: 10.1203/PDR.0b013e3182275164. PMID 21646940
- [Result] Askenazi DJ, Montesanti A, Hundley H, Koralkar R, Pawar P, Shuaib F, Liwo A, Devarajan P, Ambalavanan N. Urine biomarkers predict acute kidney injury and mortality in very low birth weight infants. J Pediatr. 2011 Dec;159(6):907-12.e1. doi: 10.1016/j.jpeds.2011.05.045. Epub 2011 Jul 23. PMID 21784446
- [Result] Auron A, Mhanna MJ. Serum creatinine in very low birth weight infants during their first days of life. J Perinatol. 2006 Dec;26(12):755-60. doi: 10.1038/sj.jp.7211604. Epub 2006 Oct 12. PMID 17036033
- [Result] Brion LP, Fleischman AR, McCarton C, Schwartz GJ. A simple estimate of glomerular filtration rate in low birth weight infants during the first year of life: noninvasive assessment of body composition and growth. J Pediatr. 1986 Oct;109(4):698-707. doi: 10.1016/s0022-3476(86)80245-1. PMID 3761090
- [Result] Carmody JB, Charlton JR. Short-term gestation, long-term risk: prematurity and chronic kidney disease. Pediatrics. 2013 Jun;131(6):1168-79. doi: 10.1542/peds.2013-0009. Epub 2013 May 13. PMID 23669525
- [Result] Carmody JB, Swanson JR, Rhone ET, Charlton JR. Recognition and reporting of AKI in very low birth weight infants. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2036-43. doi: 10.2215/CJN.05190514. Epub 2014 Oct 3. PMID 25280497
- [Result] Drukker A, Guignard JP. Renal aspects of the term and preterm infant: a selective update. Curr Opin Pediatr. 2002 Apr;14(2):175-82. doi: 10.1097/00008480-200204000-00006. PMID 11981287
- [Result] Faa G, Gerosa C, Fanni D, Nemolato S, Locci A, Cabras T, Marinelli V, Puddu M, Zaffanello M, Monga G, Fanos V. Marked interindividual variability in renal maturation of preterm infants: lessons from autopsy. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:129-33. doi: 10.3109/14767058.2010.510646. PMID 20836739
- [Result] Gadepalli SK, Selewski DT, Drongowski RA, Mychaliska GB. Acute kidney injury in congenital diaphragmatic hernia requiring extracorporeal life support: an insidious problem. J Pediatr Surg. 2011 Apr;46(4):630-635. doi: 10.1016/j.jpedsurg.2010.11.031. PMID 21496529
- [Result] Gameiro J, Branco T, Lopes JA. Artificial Intelligence in Acute Kidney Injury Risk Prediction. J Clin Med. 2020 Mar 3;9(3):678. doi: 10.3390/jcm9030678. PMID 32138284
- [Result] Genc G, Ozkaya O, Avci B, Aygun C, Kucukoduk S. Kidney injury molecule-1 as a promising biomarker for acute kidney injury in premature babies. Am J Perinatol. 2013 Mar;30(3):245-52. doi: 10.1055/s-0032-1323587. Epub 2012 Aug 8. PMID 22875659
- [Result] Guignard JP, Drukker A. Why do newborn infants have a high plasma creatinine? Pediatrics. 1999 Apr;103(4):e49. doi: 10.1542/peds.103.4.e49. PMID 10103341
- [Result] Jetton JG, Askenazi DJ. Acute kidney injury in the neonate. Clin Perinatol. 2014 Sep;41(3):487-502. doi: 10.1016/j.clp.2014.05.001. Epub 2014 Jul 22. PMID 25155722
- [Result] Jetton JG, Boohaker LJ, Sethi SK, Wazir S, Rohatgi S, Soranno DE, Chishti AS, Woroniecki R, Mammen C, Swanson JR, Sridhar S, Wong CS, Kupferman JC, Griffin RL, Askenazi DJ; Neonatal Kidney Collaborative (NKC). Incidence and outcomes of neonatal acute kidney injury (AWAKEN): a multicentre, multinational, observational cohort study. Lancet Child Adolesc Health. 2017 Nov;1(3):184-194. doi: 10.1016/S2352-4642(17)30069-X. PMID 29732396
- [Result] Jetton JG, Guillet R, Askenazi DJ, Dill L, Jacobs J, Kent AL, Selewski DT, Abitbol CL, Kaskel FJ, Mhanna MJ, Ambalavanan N, Charlton JR; Neonatal Kidney Collaborative. Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates: Design of a Retrospective Cohort Study. Front Pediatr. 2016 Jul 19;4:68. doi: 10.3389/fped.2016.00068. eCollection 2016. PMID 27486571
- [Result] Jose PA, Fildes RD, Gomez RA, Chevalier RL, Robillard JE. Neonatal renal function and physiology. Curr Opin Pediatr. 1994 Apr;6(2):172-7. doi: 10.1097/00008480-199404000-00009. PMID 8032397
- [Result] Koralkar R, Ambalavanan N, Levitan EB, McGwin G, Goldstein S, Askenazi D. Acute kidney injury reduces survival in very low birth weight infants. Pediatr Res. 2011 Apr;69(4):354-8. doi: 10.1203/PDR.0b013e31820b95ca. PMID 21178824
- [Result] Mammen C, Al Abbas A, Skippen P, Nadel H, Levine D, Collet JP, Matsell DG. Long-term risk of CKD in children surviving episodes of acute kidney injury in the intensive care unit: a prospective cohort study. Am J Kidney Dis. 2012 Apr;59(4):523-30. doi: 10.1053/j.ajkd.2011.10.048. Epub 2011 Dec 28. PMID 22206744
- [Result] Mathur NB, Agarwal HS, Maria A. Acute renal failure in neonatal sepsis. Indian J Pediatr. 2006 Jun;73(6):499-502. doi: 10.1007/BF02759894. PMID 16816511
- [Result] Miall LS, Henderson MJ, Turner AJ, Brownlee KG, Brocklebank JT, Newell SJ, Allgar VL. Plasma creatinine rises dramatically in the first 48 hours of life in preterm infants. Pediatrics. 1999 Dec;104(6):e76. doi: 10.1542/peds.104.6.e76. PMID 10586010
- [Result] Paton JB, Fisher DE, DeLannoy CW, Behrman RE. Umbilical blood flow, cardiac output, and organ blood flow in the immature baboon fetus. Am J Obstet Gynecol. 1973 Oct 15;117(4):560-6. doi: 10.1016/0002-9378(73)90122-1. No abstract available. PMID 4200569
- [Result] Rhone ET, Carmody JB, Swanson JR, Charlton JR. Nephrotoxic medication exposure in very low birth weight infants. J Matern Fetal Neonatal Med. 2014 Sep;27(14):1485-90. doi: 10.3109/14767058.2013.860522. Epub 2013 Nov 29. PMID 24168068
- [Result] Rodriguez MM, Gomez AH, Abitbol CL, Chandar JJ, Duara S, Zilleruelo GE. Histomorphometric analysis of postnatal glomerulogenesis in extremely preterm infants. Pediatr Dev Pathol. 2004 Jan-Feb;7(1):17-25. doi: 10.1007/s10024-003-3029-2. PMID 15255031
- [Result] Rudolph, A. M., Heymann, M. A., Teramo, K. A., Barrett, C. T., & Räihä, N. C. Studies on the circulation of the previable human fetus. Pediatric Research, 1971, 5.9: 452-465.
- [Result] Saint-Faust M, Boubred F, Simeoni U. Renal development and neonatal adaptation. Am J Perinatol. 2014 Oct;31(9):773-80. doi: 10.1055/s-0033-1361831. Epub 2014 Mar 12. PMID 24623338
- [Result] Salerno SN, Liao Y, Jackson W, Greenberg RG, McKinzie CJ, McCallister A, Benjamin DK, Laughon MM, Sanderson K, Clark RH, Gonzalez D. Association between Nephrotoxic Drug Combinations and Acute Kidney Injury in the Neonatal Intensive Care Unit. J Pediatr. 2021 Jan;228:213-219. doi: 10.1016/j.jpeds.2020.08.035. Epub 2020 Aug 17. PMID 32818481
- [Result] Sarafidis K, Tsepkentzi E, Agakidou E, Diamanti E, Taparkou A, Soubasi V, Papachristou F, Drossou V. Serum and urine acute kidney injury biomarkers in asphyxiated neonates. Pediatr Nephrol. 2012 Sep;27(9):1575-82. doi: 10.1007/s00467-012-2162-4. Epub 2012 Apr 25. PMID 22532328
- [Result] Sarafidis K, Tsepkentzi E, Diamanti E, Agakidou E, Taparkou A, Soubasi V, Papachristou F, Drossou V. Urine neutrophil gelatinase-associated lipocalin to predict acute kidney injury in preterm neonates. A pilot study. Pediatr Nephrol. 2014 Feb;29(2):305-10. doi: 10.1007/s00467-013-2613-6. PMID 24022367
- [Result] Sarkar S, Askenazi DJ, Jordan BK, Bhagat I, Bapuraj JR, Dechert RE, Selewski DT. Relationship between acute kidney injury and brain MRI findings in asphyxiated newborns after therapeutic hypothermia. Pediatr Res. 2014 Mar;75(3):431-5. doi: 10.1038/pr.2013.230. Epub 2013 Dec 2. PMID 24296799
- [Result] Selewski DT, Charlton JR, Jetton JG, Guillet R, Mhanna MJ, Askenazi DJ, Kent AL. Neonatal Acute Kidney Injury. Pediatrics. 2015 Aug;136(2):e463-73. doi: 10.1542/peds.2014-3819. Epub 2015 Jul 13. PMID 26169430
- [Result] Selewski DT, Jordan BK, Askenazi DJ, Dechert RE, Sarkar S. Acute kidney injury in asphyxiated newborns treated with therapeutic hypothermia. J Pediatr. 2013 Apr;162(4):725-729.e1. doi: 10.1016/j.jpeds.2012.10.002. Epub 2012 Nov 10. PMID 23149172
- [Result] Slater MB, Gruneir A, Rochon PA, Howard AW, Koren G, Parshuram CS. Identifying High-Risk Medications Associated with Acute Kidney Injury in Critically Ill Patients: A Pharmacoepidemiologic Evaluation. Paediatr Drugs. 2017 Feb;19(1):59-67. doi: 10.1007/s40272-016-0205-1. PMID 27943125
- [Result] Stoops C, Sims B, Griffin R, Askenazi DJ. Neonatal Acute Kidney Injury and the Risk of Intraventricular Hemorrhage in the Very Low Birth Weight Infant. Neonatology. 2016;110(4):307-312. doi: 10.1159/000445931. Epub 2016 Aug 5. PMID 27490643
- [Result] Stoops C, Stone S, Evans E, Dill L, Henderson T, Griffin R, Goldstein SL, Coghill C, Askenazi DJ. Baby NINJA (Nephrotoxic Injury Negated by Just-in-Time Action): Reduction of Nephrotoxic Medication-Associated Acute Kidney Injury in the Neonatal Intensive Care Unit. J Pediatr. 2019 Dec;215:223-228.e6. doi: 10.1016/j.jpeds.2019.08.046. PMID 31761141
- [Result] Sutherland MR, Gubhaju L, Moore L, Kent AL, Dahlstrom JE, Horne RS, Hoy WE, Bertram JF, Black MJ. Accelerated maturation and abnormal morphology in the preterm neonatal kidney. J Am Soc Nephrol. 2011 Jul;22(7):1365-74. doi: 10.1681/ASN.2010121266. Epub 2011 Jun 2. PMID 21636639
- [Result] Tabel Y, Elmas A, Ipek S, Karadag A, Elmas O, Ozyalin F. Urinary neutrophil gelatinase-associated lipocalin as an early biomarker for prediction of acute kidney injury in preterm infants. Am J Perinatol. 2014 Feb;31(2):167-74. doi: 10.1055/s-0033-1343770. Epub 2013 Apr 16. PMID 23592318
- [Result] Vieux R, Hascoet JM, Merdariu D, Fresson J, Guillemin F. Glomerular filtration rate reference values in very preterm infants. Pediatrics. 2010 May;125(5):e1186-92. doi: 10.1542/peds.2009-1426. Epub 2010 Apr 5. PMID 20368313
- [Result] Viswanathan S, Manyam B, Azhibekov T, Mhanna MJ. Risk factors associated with acute kidney injury in extremely low birth weight (ELBW) infants. Pediatr Nephrol. 2012 Feb;27(2):303-11. doi: 10.1007/s00467-011-1977-8. Epub 2011 Aug 3. PMID 21809002
- [Result] Yao LP, Jose PA. Developmental renal hemodynamics. Pediatr Nephrol. 1995 Oct;9(5):632-7. doi: 10.1007/BF00860962. PMID 8580030